CLINICAL TRIAL: NCT07289997
Title: Iparomlimab and Tuvonralimab Injection Combined With Apatinib and Irinotecan Hydrochloride for the Treatment of Advanced Alpha-fetoprotein-producing Gastric Cancer (AFPGC) That Progresses From First-line PD-1 Combined Chemotherapy, A Prospective, Single-arm, Phase II Clinical Study
Brief Title: Iparomlimab and Tuvonralimab Combined With Apatinib and Irinotecan Hydrochloride for the Treatment of Advanced Alpha-fetoprotein-producing Gastric Cancer (AFPGC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY011
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: AFP Gastric or Gastroesophageal Junction Adenocarcinoma; PD-1/CTLA-4; AFPGC; Immunotherapy
Keywords: immunotherapy; AFPGC; PD-1/CTLA-4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection combined with apatinib and irinotecan (Experimental): 1. Iparomlimab and Tuvonralimab Injection， 5.0mg/kg, Q3W, D1;
  2. Apatinib, 0.25g, once daily, orally; Irinotecan, 200mg/m², Q3W, D1; Combination therapy until the patient's disease progresses, or intolerable toxic and side effects occur, or until death or withdrawal of informed consent, or up to two years.
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection (QL1706)

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) — 1. Iparomlimab and Tuvonralimab Injection， 5.0mg/kg, Q3W, D1;
  2. Apatinib, 0.25g, once daily, orally; Irinotecan, 200mg/m², Q3W, D1; Combination therapy until the patient's disease progresses, or intolerable toxic and side effects occur, or until death or withdrawal of informed consent, or up to two years.

SUMMARY:
This study is a single-arm study aimed at evaluating the efficacy and safety of Iparomlimab and Tuvonralimab Injection combined with apatinib and irinotecan hydrochloride in the treatment of advanced alpha-fetoprotein gastric cancer (AFPGC) that progresses from first-line PD-1 combined with chemotherapy. The study enrolled patients with advanced gastric cancer and gastroesophageal junction cancer whose serum alpha-fetoprotein was greater than 20.0 ng/mL at the initial diagnosis and progressed after first-line PD-1 combined chemotherapy in a single center of the Fourth Hospital of Hebei Medical University. All patients underwent gastroscopy and were pathologically confirmed as Her-2 negative gastric adenocarcinoma, and had received PD-1 inhibitor treatment as the first-line treatment. Staged examinations include enhanced CT of the abdominal and pelvic cavities, plain CT scan of the chest, and color Doppler ultrasound of superficial lymph nodes. The enrolled patients received apalolitovolrelimab 5.0mg/kg, Q3W, d1; Apatinib mesylate, 0.25g, once daily; Irinotecan hydrochloride, 200mg/m², Q3W, d1. Combination therapy until the patient's disease progresses, or intolerable toxic and side effects occur, or until death or withdrawal of informed consent, or up to two years.

The primary endpoint of the study was to assess the objective response rate (ORR) of combination therapy. Secondary endpoints included progression-free survival (PFS), disease control rate (DCR), overall survival (OS), and the incidence of adverse events, etc

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study and sign the informed consent form;
2. Age≥18 years, both male and female are acceptable.
3. Unresectable，Locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction that has been diagnosed by histopathological or cytological examination, with serum alpha-fetoprotein > 20.0 ng/mL at the time of diagnosis. There is at least one measurable lesion (according to the RECIST v1.1, the long diameter of the measurable lesion on spiral CT scan is ≥10 mm or the short diameter of the enlarged lymph node is ≥15 mm; lesions that have received local treatment in the past can be used as target lesions after comfirmed progression according to the RECIST v1.1).
4. Failure of previous first-line PD-1 combined chemotherapy treatment (disease progression during or after treatment); Those who relapse within 6 months (less than 183 days) after the end of adjuvant/neoadjuvant chemotherapy (oxaliplatin combined with fluorouracil) can be included in the study, and PD-1 inhibitors need to be combined in the first-line treatment.
5. ECOG 0-1;
6. Expected survival time ≥12 weeks;
7. The functions of vital organs within 7 days before enrollment meet the following requirements (no blood components or cell growth factors are allowed to be used within 14 days before enrollment) :

   <1> Absolute neutrophil count ≥1.5×109/L; <2> platelet count ≥80×109/L; <3>Hemoglobin ≥9g/dL; <4>Total bilirubin < 1.5 times ULN; <5>ALT and AST < 2.5 times ULN (< 5 times ULN in patients with liver metastasis); <6> serum creatinine ≤1 times ULN; <7>The endogenous creatinine clearance rate ≥ 50ml/min.
8. Women of childbearing age should take effective contraceptive measures.
9. Good compliance and cooperation with follow-up visits.

Exclusion Criteria:

1. Inability to comply with the research plan or procedures;
2. It is known to be in a HER2-positive state;
3. Gastric cancer known to be squamous cell carcinoma, undifferentiated carcinoma or other tissue types, or adenocarcinoma mixed with other tissue types of gastric cancer;
4. The patient currently has any diseases or conditions that affect the absorption of the drug;
5. Combined with severe cardiovascular diseases, such as uncontrollable heart failure, coronary heart disease, arrhythmia, uncontrollable hypertension, etc.
6. Patients with active brain metastases. Patients with asymptomatic brain metastases who have not received prior treatment and whose total number of brain metastases is ≤3 and the longest diameter is < 1cm can be enrolled. Patients who have previously received treatment for brain metastases can be enrolled if they are clinically stable, have no evidence of new or expanded brain metastases, and have not used steroids for ≥14 days before the study intervention.
7. Known to be allergic to the drug used in this test;
8. Previously received immune checkpoint inhibitors other than anti-PD-1 /PD-L1 antibodies or other drugs/antibodies acting on T-cell co-stimulation or checkpoint pathways;
9. Significant clinically significant bleeding symptoms or a clear bleeding tendency occurred within 3 months before enrollment; Gastrointestinal perforation and/or gastrointestinal fistula occurred within 6 months before enrollment; Arterial/venous thrombotic events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
10. Clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or hepatitis C (previous history of hepatitis B virus infection regardless of drug control, hepatitis B virus DNA≥1×104 copies /mL or 2000 IU/ml);
11. Known history of primary immunodeficiency or active pulmonary tuberculosis;
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
13. There is a known history of human immunodeficiency virus (HIV) infection (i.e., HIV antibody positive);
14. Significant malnutrition (weight loss of 5% within one month of signing the informed consent form or 15% within three months, or a reduction of half or more in food intake within one week), except for more than four weeks after the correction of malnutrition before the administration of the first dose of the study drug;
15. History of other primary malignant tumors, excluding:

    <1>Malignant tumors that achieved complete remission for at least 2 years before enrollment and did not require additional treatment during the study period; <2>Non-melanoma skin cancer or malignant freckle-like nevus that has been fully treated and has no evidence of disease recurrence; <3>Carcinoma in situ that has received adequate treatment and has no evidence of disease recurrence.
16. Female patients who are pregnant or breastfeeding;
17. According to the researcher's judgment, those with concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study;
18. The researchers considered patients unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24months
  The objective response rate (ORR), which is the proportion of patients with complete response and partial response as assessed according to the RECIST1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 36month
  The period from the start of treatment to disease progression, death from any cause, or the end of follow-up, whichever occurs first
Overall survival (OS) | 48months
  The time from the start of treatment to death due to any cause or the end of follow-up
Disease control rate (DCR) | 24months
  Disease control rate (DCR) : It refers to the proportion of patients who achieved PR、CR and SD after treatment. DCR=CR+PR+SD
Adverse Events（AEs） | 36months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No